CLINICAL TRIAL: NCT04974697
Title: Evaluation of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6435
Record Dates: First submitted 2021-07-19; First posted 2021-07-23 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Subjects will be masked to the study lens to help reduce potential bias. Subjects will be unaware of the identity of the investigational product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- JJVC Investigational Multifocal Toric Contact Lens (Experimental): Eligible subjects that are adapted contact lens wearers with presbyopia, ametropia (hyperopia or myopia) and astigmatism will be dispensed the study lens in a bilateral fashion.
  Interventions: Device: JJVC Investigational Multifocal Toric Contact Lens

INTERVENTIONS:
Device: JJVC Investigational Multifocal Toric Contact Lens — TEST

SUMMARY:
The study is a bilateral, single-masked, single-arm, 4-visit dispensing study. There will be one study treatment, with the subject being dispensed lenses for 6 to 8 days, then lens power will be optimized (if necessary) and dispensed for a further 2 weeks to assess the clinical performance of investigational multifocal toric contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be at least 40 and not more than 70 years of age at the time of screening.
  4. Own a wearable pair of spectacles if required for their distance vision.
  5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks).
  6. Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
  7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +3.75 D.
  8. The subject's refractive cylinder must be -1.00 D to -1.50 D in each eye, with the cylinder axes in the range of 90°±30°.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
  10. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use systemic medications that may interfere with contact lens wear or cause blurred vision.
  4. Currently use ocular medication (with the exception of rewetting drops).
  5. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
  6. Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, cataract surgery, retinal surgery, etc.).
  7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.
  8. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  10. Have a history of amblyopia or strabismus, by self-report.
  11. Have a history of herpetic keratitis, by self-report.
  12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (8):
- United States (8):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - VRC-West, Jacksonville, Florida
  - Maitland Vision Center, Maitland, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Township, Michigan
  - Eye Associates of New York, New York, New York
  - Sacco Eye Group, Vestal, New York
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 95 subjects were enrolled into this study. Of those enrolled, 86 were dispensed study lenses, while 9 subjects failed to meet all eligibility criteria. Of those dispensed, 84 completed the study while 2 subjects were discontinued.
Groups:
- Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker: Subjects that wore the multifocal toric Contact Lens in senofilcon A (C3) with UV/HEV blocker during any point of the study.
Period: Overall Study
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Started | 86
Completed | 84
Not Completed | 2
Not completed — Unsatisfactory lens fitting due to test article | 1
Not completed — Lens discomfort | 1

BASELINE CHARACTERISTICS:
Population: All Subjects dispensed a study lens.
Groups:
- Myope: subjects were classified as Myopic if the distance spherical component of their refractive error was in the range of -1.25 D to -3.75 D
- Hyperope: subjects were classified as Hyperopic if the distance spherical component of their refractive error was in the range of +1.25 D to +3.75 D
- Total: Total of all reporting groups
Arm/Group | Myope | Hyperope | Total
Number analyzed (Participants) | 48 | 38 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (6.28) | 56.7 (7.36) | 52.2 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 43 | 32 | 75
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 38 | 86

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20),where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: Subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker: Subject that wore the multifocal toric contact lens in senofilcon A (C3) with UV/HEV blocker throughout the entire duration of the study. The average CLUE vision score for each sphere stratum (Hyperope and Myope) was reported.
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Number analyzed (Participants) | 83
Units on a Scale
  Myope: number analyzed (Participants) | 48
  Myope | 58.37 (21.586)
  Hyperope: number analyzed (Participants) | 35
  Hyperope | 53.53 (21.160)
Statistical Analysis 1: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; It was calculated using a 2-sided one sample means t-test with a family wise type I error rate of 5% and at least 80% statistical power, that 22 subjects were required to test superiority for myope; Test type: Superiority — The superiority of the test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold 40 points for myope; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 58.1, 95% CI 2-sided [50.9 to 65.4], Standard Error of Mean 3.37
Statistical Analysis 2: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; It was calculated using a 2-sided one sample means t-test with a family wise type I error rate of 5% and at least 80% statistical power, that 18 subjects were required to test superiority for hyperope; Test type: Superiority — The superiority of the test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold 32 points for hyperope; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 55.0, 95% CI 2-sided [47.2 to 62.8], Standard Error of Mean 3.70

2. Primary Outcome: LogMAR Visual Acuity
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 m),intermediate (64 cm) and near (40 cm) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. The room illuminance was required to be between 7.3 and 7.9 EV (394-597 lux). For Distance (4 m), the acceptable range for the chart luminance was 10.5-10.7 EV (181-208 cd/m2). For Intermediate (64cm) and Near (40cm), the acceptable range for the chart luminance 10.8-11.1 EV (223-274 cd/m2). Letter by-letter results calculated the visual performance score for each chart read. A logMAR score closer to zero, or below zero, indicates a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20. Hyperopes and myopes were combined based on historical data for subjects in this study with regard to visual performance logMAR.
Time Frame: 2-Week Follow-up
Population: Subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Number analyzed (Participants) | 83
LogMAR
  Distance (4M) | -0.12 (0.083)
  Intermediate (64 cm) | -0.05 (0.089)
  Near (40 cm) | 0.06 (0.125)
Statistical Analysis 1: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; It was calculated by using a 2-sided one sample mean t-test with a family wise type I error rate of 5% and at least 80% statistical power , 42 subjects were required to test superiority for distance (4m); Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold 0.00 logMAR for Distance; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = -0.129, 95% CI 2-sided [-0.167 to -0.091], Standard Error of Mean 0.0166
Statistical Analysis 2: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; It was calculated by using a 2-sided one sample mean t-test with a family wise type I error rate of 5% and at least 80% statistical power , 7 subjects were required to test superiority for intermediate (64 cm); Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold +0.17 logMAR for Intermediate; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = -0.046, 95% CI 2-sided [-0.084 to -0.008], Standard Error of Mean 0.0166
Statistical Analysis 3: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; It was calculated by using a 2-sided one sample mean t-test with a family wise type I error rate of 5% and at least 80% statistical power , 36 subjects were required to test superiority for near (40 cm); Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold +0.17 logMAR for Near; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 0.067, 95% CI 2-sided [0.029 to 0.105], Standard Error of Mean 0.0166

3. Secondary Outcome: Change From Baseline CLUE Vision Score
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The change from baseline was calculated as the 2 week follow-up scores minus baseline scores. Change from baseline scores range from -120 to 120, where higher change from baseline scores indicate better performance. The average change from baseline was reported.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker: Subject that wore the multifocal toric contact lens in senofilcon A (C3) with UV/HEV blocker throughout the entire duration of the study.
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Number analyzed (Participants) | 83
Units on a Scale
  Myope: number analyzed (Participants) | 48
  Myope | 8.40 (18.163)
  Hyperope: number analyzed (Participants) | 35
  Hyperope | 5.03 (18.799)
Statistical Analysis 1: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — The non-inferiority of the test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold -5 points for myope; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 8.4, 95% CI 2-sided [3.1 to 13.7], Standard Error of Mean 2.66
Statistical Analysis 2: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — The non-inferiority of the test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold -5 points for hyperope; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 5.0, 95% CI 2-sided [-1.2 to 11.2], Standard Error of Mean 3.12

4. Secondary Outcome: Change From Baseline CLUE Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The change from baseline was calculated as the 2- week follow-up scores minus baseline scores. Change from baseline scores range from -120 to 120, where higher change from baseline scores indicate better performance. The average change from baseline was reported.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Number analyzed (Participants) | 83
Units on a Scale
  Myope: number analyzed (Participants) | 48
  Myope | 6.85 (22.912)
  Hyperope: number analyzed (Participants) | 35
  Hyperope | 3.30 (25.123)
Statistical Analysis 1: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 6.9, 95% CI 2-sided [0.0 to 13.7], Standard Error of Mean 3.44
Statistical Analysis 2: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 3.3, 95% CI 2-sided [-4.7 to 11.3], Standard Error of Mean 4.03

5. Secondary Outcome: Change From Baseline CLUE Handling Score
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18- 65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The change from baseline was calculated as the 2- week follow-up scores minus baseline scores. Change from baseline scores range from -120 to 120, where higher change from baseline scores indicate better performance. The average change from baseline was reported.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
Number analyzed (Participants) | 83
Units on a Scale
  Myope: number analyzed (Participants) | 48
  Myope | 11.22 (22.261)
  Hyperope: number analyzed (Participants) | 35
  Hyperope | 10.02 (20.553)
Statistical Analysis 1: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 11.2, 95% CI 2-sided [5.0 to 17.4], Standard Error of Mean 3.11
Statistical Analysis 2: Comparison: Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker; The study was only powered for the primary endpoint; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 10.0, 95% CI 2-sided [2.8 to 17.3], Standard Error of Mean 3.64

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 3 weeks per subject.
Arm/Group | Multifocal Toric Contact Lens in Senofilcon A (C3) With UV/HEV Blocker
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT04974697/Prot_SAP_000.pdf